CLINICAL TRIAL: NCT03827395
Title: A Phase 1, Double-Blinded, Placebo Controlled, Clinical Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of HEV-239 (Hecolin(R)) in a Healthy US Adult Population
Brief Title: Safety Study of Hepatitis E Vaccine (HEV239)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-0108; HHSN272201300018I
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-10-16

CONDITIONS: Hepatitis E; Immunisation
Keywords: Adult; Healthy; Hecolin; Hepatitis E; HEV239; Immunogenicity; Placebo; Population; Reactogenicity; Route; Safety; Vaccine
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEV-239 (Experimental): 0.5 mL of HEV-239 administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180. N=20
  Interventions: Biological: HEV 239
- Placebo (Placebo Comparator): 0.5 mL of HEV-239 placebo administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180. N=5
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HEV 239 — Hepatitis E vaccine against HEV genotypes 1 and 4. The HEV 239 vaccine is a 26 kDa recombinant polypeptide corresponding to amino acid residues 368-606 of the capsid protein of a genotype 1 HEV strain. The vaccine is expressed in Escherichia coli (E. coli) and vaccine doses contain 30 µg of the purified antigen in 0.5 mL buffered saline adsorbed to 0.8 mg aluminium hydroxide.
  Arms: HEV-239
Other: Placebo — 0.9% Sodium Chloride Injection, USP (Normal Saline) is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection (WFI). Each mL contains sodium chloride 9 mg and may contain HCl or NaOH for pH adjustment (pH 5.3 [4.5 - 7.0]).
  Arms: Placebo

SUMMARY:
This is a Phase I double-blind, randomized, placebo controlled trial (1:4 ratio of placebo to vaccine) of Hepatitis E virus vaccine containing a 239 amino acid subfragment of Hecolin(R) (HEV-239) in 25 US males and non-pregnant females ages 18 - 45 (inclusive) to assess the safety, reactogenicity, and immunogenicity of HEV-239. Subjects will receive 3 doses of study product on Days 1, 29, and 180. Subjects will remain in the study for up to 13 months (including screening). The study duration will be approximately 15 months. Subjects will be observed for 30 minutes after vaccination. The occurrence of solicited injection site and systemic reactogenicity events will be measured from the time of study vaccination through Day 8 after each vaccination. These will be ascertained through use of an electronic memory (e-memory) aid, a telephone call on day 4 after each dose of vaccine, a Day 8 clinic visit, and potentially at the Day 15 clinic visit after each dose of vaccine. Unsolicited adverse events will be collected from vaccination through Day 29 after each vaccination. Serious adverse events will be collected from the time of the first study vaccination through the last study visit (Day 360). The study includes multiple phlebotomy time points for immunogenicity and blood collection for future use at visit 1 and Days 8, 15, and 29 after each vaccination. The durability of the immune response and future use collection will be assessed at 5 months after the first boost (Day 180) and at 6 months after the second boost (Day 360). The primary objectives of the study are to; 1) assess the safety and reactogenicity of HEV-239 following delivery of each vaccine dose; and 2) assess the number of subjects with > / = 4 fold rise in Hepatitis E virus (HEV) immunoglobulin G (IgG) at any time after vaccination.

DETAILED DESCRIPTION:
This is a Phase I double-blind, randomized, placebo controlled trial (1:4 ratio of placebo to vaccine) of Hepatitis E virus vaccine containing a 239 amino acid subfragment of Hecolin(R) (HEV-239) in 25 US males and non-pregnant females ages 18 - 45 (inclusive) to assess the safety, reactogenicity, and immunogenicity of HEV-239. Subjects will receive 3 doses of study product on Days 1, 29, and 180. Subjects will remain in the study for up to 13 months (including screening). The study duration will be approximately 15 months. Subjects will be observed for 30 minutes after vaccination. The occurrence of solicited injection site and systemic reactogenicity events will be measured from the time of study vaccination through Day 8 after each vaccination. These will be ascertained through use of an electronic memory (e-memory) aid, a telephone call on day 4 after each dose of vaccine, a Day 8 clinic visit, and potentially at the Day 15 clinic visit after each dose of vaccine. Unsolicited adverse events will be collected from vaccination through Day 29 after each vaccination. Serious adverse events will be collected from the time of the first study vaccination through the last study visit (Day 360). The study includes multiple phlebotomy time points for immunogenicity and blood collection for future use at visit 1 and Days 8, 15, and 29 after each vaccination. The durability of the immune response and future use collection will be assessed at 5 months after the first boost (Day 180) and at 6 months after the second boost (Day 360). The primary objectives of the study are to; 1) Assess the safety and reactogenicity of HEV-239 following delivery of each vaccine dose; and 2) Assess the number of subjects with > / = 4 fold rise in Hepatitis E virus (HEV) immunoglobulin G (IgG) at any time after vaccination. The secondary objectives are to; 1) Assess the number of subjects with HEV immunoglobulin M (IgM) seroconversion at any time after vaccination; 2) Assess the number of subjects with HEV IgG seroconversion at any time after vaccination; and 3) Assess the HEV IgG geometric mean concentrations (GMCs) at any time after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent.
2. Subject must be able to comprehend and willing to comply with all study visits and procedures (up to 13 months from enrollment).
3. Subject must be a man or a non-pregnant woman* aged 18-45 years (inclusive).

   *Females of childbearing potential must have a negative serum human chorionic gonadotropin (beta-HCG) pregnancy test at screening and negative urine beta-HCG pregnancy test within 24 hours prior to (each) vaccination.
4. Subject must be in good general health as determined by medical history, vital signs*, body mass index (BMI)**, physical examination, and clinical judgment of the investigator.

   *Oral temp < 38.0 Degrees Celsius /100.4 Degrees Fahrenheit; pulse 51 to 100 bpm; systolic blood pressure 90 to 140 mm Hg, and diastolic blood pressure 55 to 90 mm Hg.

   **BMI > / = 18.5 and < 35 kg/m^2.
5. Subject's screening laboratory values*,** must be within site normal limits*** within 28 days of enrollment.

   *Screening labs will include: White blood cell (WBC) count; Hemoglobin (HgB); Platelets; Absolute neutrophil count (ANC); Absolute eosinophil count (AEC); Creatinine; Glucose (random, must be < 140); Alanine Aminotransferase (ALT); HIV 1/2 antibody/antigen test, Hepatitis B surface antigen (HBsAg), and Hepatitis C virus (HCV) antibody.

   **Minor abnormalities are considered acceptable if not clinically significant (e.g., Mean Corpuscular Volume (MCV)). Repeating the screening tests once is permitted for out-of-range values provided there is an alternative explanation for the out-of-range value. The alternative explanation for the out-of-range value should be documented in the subject's source documents.

   ***Creatinine, glucose, and ALT values lower than the normal range may be acceptable if the PI or a designated licensed clinician determines that these laboratory findings are not clinically significant. The HIV 1/2 antibody/antigen test, Hepatitis B surface antigen (HBsAg), and Hepatitis C virus (HCV) antibody must be non-reactive.
6. Subject's Hepatitis E Virus (HEV) - specific Immunoglobulin G (IgG) and Immunoglobulin M (IgM) are negative by ELISA at screening.
7. Subject agrees to not to participate in another clinical trial during the study period.
8. Subject agrees not to donate blood from screening through Day 270.
9. Female subjects must be of non-childbearing potential* OR must use an acceptable method of contraception** from 28 days before prime vaccination until at least 3 months after the last vaccination.

   *Surgically sterile via tubal ligation, bilateral oophorectomy, hysterectomy or postmenopausal for > / = 1 year.

   **Abstinence (defined as refraining from heterosexual intercourse), monogamous relationship with vasectomized partner, barrier methods such as male or female condoms with spermicide or diaphragms with spermicide, intrauterine devices, and licensed hormonal methods (such as birth control pills, skin patches, Implanon(R), Nexplanon(R), DepoProvera(R), or NuvaRing(R)).
10. Male subjects must be surgically sterile via vasectomy OR must use an acceptable method of contraception* from prime vaccination until at least 3 months after the last boost vaccination.

    * Abstinence (defined as refraining from heterosexual intercourse), or condoms with spermicide.
11. Subjects must have consistent access to the internet to perform electronic data entry.

Exclusion Criteria:

1. Has a previous HEV infection or chronic liver disease.
2. Has received any experimental agent* within 30 days prior to first vaccination, or the expected recipient of any experimental agent during this trial-reporting period.

   *Including vaccines, drugs, biologics, devices, and/or blood products.
3. Female subject is pregnant (or has a positive pregnancy test prior to vaccination) or breast feeding, or planning to become pregnant within 3 months after the last boost vaccination.
4. Fever (> / = 38.0 Degrees Celsius / 100.4 Degrees Fahrenheit) or other acute illness within 3 days prior to first vaccination.
5. Infection requiring systemic antibiotics or antiviral treatment within the 7 days prior to first vaccination.
6. Has a positive urine drug screen for amphetamines*, cocaine, opiates, or phencyclidine.

   *Prescription amphetamines are not exclusionary.
7. Chronic, clinically significant medical or psychiatric conditions* that, in the opinion of the investigator, may pose additional risk to the subject if she/he participates in the study.

   *Permissible conditions include but are not limited to mild, well-controlled asthma, well-controlled depression, well-controlled anxiety, seasonal allergies, and well-controlled hypertension.
8. Receipt of immunosuppressive drugs*,**,*** or biologic agents within the 30 days prior to enrollment.

   *This includes use of oral or parental prednisone. This also includes allergy desensitization injections from 14 days prior to each vaccination through 14 days after each vaccination. The use of topical steroids for mild uncomplicated dermatitis permissible after therapy is completed. Over-the-counter (OTC) corticosteroid nasal sprays for allergic rhinitis are permissible. The use of low or moderate dose inhaled steroids is permissible. Doses are defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.

   **Receipt of systemic, prescription medications for the treatment of chronic medical conditions or variations of normal physiologic functions may be permissible if, in the opinion of the investigator, they are used for conditions that are not clinically significant and would not impact the safety of the subject or the safety and immunogenicity outcomes of the protocol.

   ***Use of systemic, over-the-counter medications and PRN systemic, prescription medication may be allowed if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of immunogenicity/reactogenicity.
9. Has known neoplastic disease* anticancer therapy, or radiation therapy within 3 years prior to first study vaccination.

   *Excluding non-melanoma skin cancer, such as squamous cell skin cancer or basal cell skin cancer, cured by surgical excision.
10. Has a history of any hematologic malignancy at any time.
11. Has a known or suspected congenital or acquired disease that impairs the immune system, including functional asplenia or immunosuppression as a result of underlying illness or treatment.
12. Has prior organ and/or stem cell transplant.
13. Has a history of abuse of alcohol or drugs that, in the opinion of the investigator, may interfere with the subject's ability to comply with the protocol.
14. Has behavioral or cognitive impairment or psychiatric conditions that, in the opinion of the investigator, may interfere with the subject's ability to participate in the trial.
15. Has received blood products or immunoglobulin within six months prior to vaccination.
16. Travel to Asia, the Middle East, Africa, or Central America or to an area with an active Hepatitis E outbreak* within the last 90 days or intention to travel to such areas during the study.

    *Outbreaks within the last 3 years.
17. Receipt of any inactivated vaccine from 2 weeks prior to each vaccination through 2 weeks after each vaccination.
18. Receipt of any live vaccine from 4 weeks prior to each vaccination through 4 weeks after each vaccination.
19. Known hypersensitivity or allergy to aluminum, any component of the vaccine, or other serious adverse reactions to vaccines or vaccine products.
20. Subject who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study.
21. Any condition that, in the opinion of the investigator, might interfere with assessing the study objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kao CM, Rostad CA, Nolan LE, Peters E, Kleinhenz J, Sherman JD, Tippett A, Shih JWK, Yildirim I, Agbakoba V, Beresnev T, Ballou C, Kamidani S, Karmali V, Natrajan M, Scherer EM, Rouphael N, Anderson EJ. A Phase 1, Double-Blinded, Placebo-Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of HEV-239 (Hecolin) Vaccine in Healthy US Adults. J Infect Dis. 2024 Nov 15;230(5):1093-1101. doi: 10.1093/infdis/jiae148. PMID 38536442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 18 and 45 years old, inclusively. They were recruited from the community at large around the clinical site. Participants were enrolled between 12APR2019 and 24JUL2019.
Groups:
- HEV-239: 0.5 mL of HEV-239 administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180.
  HEV 239: Hepatitis E vaccine against HEV genotypes 1 and 4. The HEV 239 vaccine is a 26 kDa recombinant polypeptide corresponding to amino acid residues 368-606 of the capsid protein of a genotype 1 HEV strain. The vaccine is expressed in Escherichia coli (E. coli) and vaccine doses contain 30 µg of the purified antigen in 0.5 mL buffered saline adsorbed to 0.8 mg aluminium hydroxide.
- Placebo: 0.5 mL of HEV-239 placebo administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180.
  Placebo: 0.9% Sodium Chloride Injection, USP (Normal Saline) is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection (WFI). Each mL contains sodium chloride 9 mg and may contain HCl or NaOH for pH adjustment (pH 5.3 [4.5 - 7.0]).
Period: Overall Study
Arm/Group | HEV-239 | Placebo
Started | 20 | 5
Completed | 17 | 3
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Became ineligible after enrollment | 1 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who were enrolled in the study
Groups:
- HEV-239: 0.5 mL of HEV-239 administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180.
- Placebo: 0.5 mL of HEV-239 placebo administered intramuscularly into the deltoid muscle as a single injection on Days 1, 29, and 180.
- Total: Total of all reporting groups
Arm/Group | HEV-239 | Placebo | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 5 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (6.7) | 32.8 (7.9) | 30.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 15 | 3 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactogenicity Events
Description: Injection site Adverse Events (AEs) solicited on an e-memory aid available to participants included: pain, tenderness, pruritis/itching, ecchymosis/bruising, induration/swelling (functional grade based on interference with daily activities). Ecchymosis/bruising (any measured value >/= 25mm), induration/swelling (any measured value >/= 25mm), and erythema/redness (any measured value >/= 25mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following vaccination.
Time Frame: Post Dose 1 (Day 1 through Day 8), Post Dose 2 (Day 29 through Day 36), Post Dose 3 (Day 180 through Day 187)
Population: The Safety Analysis population includes all participants who received at least one study vaccination and for whom data at the corresponding time point exists.
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants
  Post Dose 1 | 11 | 3
  Post Dose 2: number analyzed (Participants) | 20 | 3
  Post Dose 2 | 17 | 1
  Post Dose 3: number analyzed (Participants) | 19 | 3
  Post Dose 3 | 9 | 1
  Post Any Dose | 19 | 3

2. Primary Outcome: Number of Participants With Solicited Systemic Reactogenicity Events
Description: Systemic AEs solicited on an e-memory aid provided to participants included: feverishness, fatigue, malaise, myalgia, arthralgia, headache, nausea, vomiting, and elevated oral temperature (38.0 degrees Celsius/100.4 degrees Fahrenheit or greater). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following vaccination.
Time Frame: Post Dose 1 (Day 1 through Day 8), Post Dose 2 (Day 29 through Day 36), Post Dose 3 (Day 180 through Day 187)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants
  Post Dose 1 | 11 | 3
  Post Dose 2: number analyzed (Participants) | 20 | 3
  Post Dose 2 | 12 | 1
  Post Dose 3: number analyzed (Participants) | 19 | 3
  Post Dose 3 | 7 | 1
  Post Any Dose | 17 | 4

3. Primary Outcome: Number of Participants With Vaccine-related Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Unsolicited AEs that were deemed vaccine-related were collected from participants from the time of vaccination through Day 29 after each study vaccination.
Time Frame: Post Dose 1 (Day 1 through Day 29), Post Dose 2 (Day 29 through Day 57), Post Dose 3 (Day 180 through Day 208)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events (AEs) - Chemistry
Description: Chemistry parameters included: alanine aminotransferase (ALT) and creatinine. Thresholds for adverse events were considered as ALT 30 U/L or greater (female) or 47 U/L or greater (male); creatinine 1.11 mg/dL or greater (female) or 1.36 mg/dL or greater (male).
Time Frame: Baseline, Post Dose 1 (Day 8), Post Dose 2 (Day 36), Post Dose 3 (Day 187)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events (AEs) - Hematology
Description: Hematology parameters included: hemoglobin, platelets, absolute neutrophil count (ANC), absolute eosinophil count (AEC), and white blood cells (WBC). Thresholds for adverse events were considered as hemoglobin 11.0 g/dL or greater (female) or 12.0 g/dL or greater (male); WBC increase 10.9 thousand/uL or greater; WBC decrease 3.7 thousand/uL or less; ANC decrease 1499 cells/uL or less; AEC increase 501 cells/uL or greater; platelet decrease 139 thousand/uL or less.
Time Frame: Baseline, Post Dose 1 (Day 8), Post Dose 2 (Day 36), Post Dose 3 (Day 187)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants
  Baseline: None | 20 | 5
  Baseline: Mild/Grade 1 | 0 | 0
  Baseline: Moderate/Grade 2 | 0 | 0
  Baseline: Severe/Grade 3 | 0 | 0
  Baseline: Missing | 0 | 0
  Post Dose 1: None | 20 | 5
  Post Dose 1: Mild/Grade 1 | 0 | 0
  Post Dose 1: Moderate/Grade 2 | 0 | 0
  Post Dose 1: Severe/Grade 3 | 0 | 0
  Post Dose 1: Missing | 0 | 0
  Post Dose 2: None | 19 | 3
  Post Dose 2: Mild/Grade 1 | 0 | 0
  Post Dose 2: Moderate/Grade 2 | 1 | 0
  Post Dose 2: Severe/Grade 3 | 0 | 0
  Post Dose 2: Missing | 0 | 2
  Post Dose 3: number analyzed (Participants) | 19 | 3
  Post Dose 3: None | 17 | 3
  Post Dose 3: Mild/Grade 1 | 0 | 0
  Post Dose 3: Moderate/Grade 2 | 1 | 0
  Post Dose 3: Severe/Grade 3 | 0 | 0
  Post Dose 3: Missing | 1 | 0

6. Primary Outcome: Number of Participants With Vaccine-related Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect; or any important medical event that may not result in death, be life-threatening, or require hospitalizations, that may be considered serious when, based on appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 360
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Participants | 0 | 0

7. Primary Outcome: Percentage of Participants Showing >/=4-fold Rise in Serum Hepatitis E Virus Immunoglobulin G (IgG) Concentration
Description: Blood was collected for IgG assay which was conducted with HEV as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean fold rise was calculated for each study arm from the available results at Day 8 and Day 15 post first study vaccination, Day 29 prior to second study vaccination, Day 36, Day 43, Day 57, Day 180 prior to third study vaccination, Day 187, Day 194, Day 208 and Day 360. A 4-fold rise was defined as a HEV IgG >/=0.154 Wu/mL in a participant that was HEV seronegative at Day 1.
Time Frame: Day 8, Day 15, Day 29 (Dose 2), Day 36, Day 43, Day 57, Day 180 (Dose 3), Day 187, Day 194, Day 208, Day 360
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination blood sample for immunogenicity testing for which valid results were reported at the corresponding time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
percentage of participants
  Day 8 | 0 [0 to 17] | 0 [0 to 52]
  Day 15 | 65 [41 to 85] | 0 [0 to 52]
  Day 29 (Dose 2) | 100 [83 to 100] | 0 [0 to 52]
  Day 36: number analyzed (Participants) | 20 | 3
  Day 36 | 100 [83 to 100] | 0 [0 to 71]
  Day 43: number analyzed (Participants) | 19 | 3
  Day 43 | 100 [82 to 100] | 0 [0 to 71]
  Day 57 | 100 [83 to 100] | 0 [0 to 52]
  Day 180 (Dose 3): number analyzed (Participants) | 19 | 5
  Day 180 (Dose 3) | 100 [82 to 100] | 0 [0 to 52]
  Day 187: number analyzed (Participants) | 18 | 3
  Day 187 | 100 [81 to 100] | 0 [0 to 71]
  Day 194: number analyzed (Participants) | 18 | 3
  Day 194 | 100 [81 to 100] | 0 [0 to 71]
  Day 208: number analyzed (Participants) | 19 | 3
  Day 208 | 100 [82 to 100] | 0 [0 to 71]
  Day 360: number analyzed (Participants) | 17 | 3
  Day 360 | 100 [80 to 100] | 0 [0 to 71]

8. Secondary Outcome: Percentage of Participants With Hepatitis E Virus Immunoglobulin M (IgM) Seroconversion
Description: Blood was collected for the IgM assay conducted with HEV as the antigen. Each sample was tested in duplicate per the laboratory's standard operating procedure and retested in duplicate if a result was borderline (A / C.O. = 0.9-1.1). If any replicate was seropositive [A/C.O. >1.1 as defined by the Wantai HEV-IgM enzyme-linked immunosorbent assay (ELISA) package insert] the sample's result was positive. If no replicates were positive the sample's result was negative. Seroconversion was defined as a change from a seronegative result to a seropositive result.
Time Frame: Day 8, Day 15, Day 29 (Dose 2), Day 36, Day 43, Day 57, Day 180 (Dose 3), Day 187, Day 194, Day 208, Day 360
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
percentage of participants
  Day 8 | 0 [0 to 17] | 0 [0 to 52]
  Day 15 | 0 [0 to 17] | 0 [0 to 52]
  Day 29 (Dose 2) | 15 [3 to 38] | 0 [0 to 52]
  Day 36: number analyzed (Participants) | 20 | 3
  Day 36 | 15 [3 to 38] | 0 [0 to 71]
  Day 43: number analyzed (Participants) | 19 | 3
  Day 43 | 16 [3 to 40] | 0 [0 to 71]
  Day 57 | 10 [1 to 32] | 0 [0 to 52]
  Day 180 (Dose 3): number analyzed (Participants) | 19 | 5
  Day 180 (Dose 3) | 0 [0 to 18] | 0 [0 to 52]
  Day 187: number analyzed (Participants) | 18 | 3
  Day 187 | 0 [0 to 19] | 0 [0 to 71]
  Day 194: number analyzed (Participants) | 18 | 3
  Day 194 | 0 [0 to 19] | 0 [0 to 71]
  Day 208: number analyzed (Participants) | 19 | 3
  Day 208 | 0 [0 to 18] | 0 [0 to 71]
  Day 360: number analyzed (Participants) | 17 | 3
  Day 360 | 0 [0 to 20] | 0 [0 to 71]

9. Secondary Outcome: Percentage of Participants With Hepatitis E Virus IgG Seroconversion
Description: Blood was collected for the IgG assay conducted with HEV as the antigen. Each sample was tested in duplicate per the laboratory's standard operating procedure and retested in duplicate if a result was borderline (A / C.O. = 0.9-1.1). If any replicate was seropositive (A/C.O. >1.1 as defined by the Wantai HEV-IgG ELISA package insert) the sample's result was positive. If no replicates were positive the sample's result was negative. Seroconversion was defined as a change from a seronegative result to a seropositive result.
Time Frame: Day 8, Day 15, Day 29 (Dose 2), Day 36, Day 43, Day 57, Day 180 (Dose 3), Day 187, Day 194, Day 208, Day 360
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
percentage of participants
  Day 8 | 0 [0 to 17] | 0 [0 to 52]
  Day 15 | 60 [36 to 81] | 0 [0 to 52]
  Day 29 (Dose 2) | 100 [83 to 100] | 0 [0 to 52]
  Day 36: number analyzed (Participants) | 20 | 3
  Day 36 | 100 [83 to 100] | 0 [0 to 71]
  Day 43: number analyzed (Participants) | 19 | 3
  Day 43 | 100 [82 to 100] | 0 [0 to 71]
  Day 57 | 100 [83 to 100] | 0 [0 to 52]
  Day 180 (Dose 3): number analyzed (Participants) | 19 | 5
  Day 180 (Dose 3) | 100 [82 to 100] | 0 [0 to 52]
  Day 187: number analyzed (Participants) | 18 | 3
  Day 187 | 100 [81 to 100] | 0 [0 to 71]
  Day 194: number analyzed (Participants) | 18 | 3
  Day 194 | 100 [81 to 100] | 0 [0 to 71]
  Day 208: number analyzed (Participants) | 19 | 3
  Day 208 | 100 [82 to 100] | 0 [0 to 71]
  Day 360: number analyzed (Participants) | 17 | 3
  Day 360 | 100 [80 to 100] | 0 [0 to 71]

10. Secondary Outcome: Geometric Mean Concentrations (GMC) of Hepatitis E Virus IgG
Description: Blood was collected for IgG assay which was conducted with HEV as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean concentration (Wu/mL) was calculated for each study arm from the available results at each timepoint.
Time Frame: Day 1 (Dose 1), Day 8, Day 15, Day 29 (Dose 2), Day 36, Day 43, Day 57, Day 180 (Dose 3), Day 187, Day 194, Day 208, Day 360
Population: as for outcome 7
Measure: Geometric Mean (Full Range); unit: Wu/mL
Arm/Group | HEV-239 | Placebo
Number analyzed (Participants) | 20 | 5
Wu/mL
  Day 1 (Dose 1) | 0.0385 [0.0385 to 0.0385] | 0.0385 [0.0385 to 0.0385]
  Day 8 | 0.0385 [0.0385 to 0.0385] | 0.0385 [0.0385 to 0.0385]
  Day 15 | 0.24999 [0.0385 to 1.4405] | 0.0385 [0.0385 to 0.0385]
  Day 29 (Dose 2) | 1.44483 [0.2175 to 8.9019] | 0.0385 [0.0385 to 0.0385]
  Day 36: number analyzed (Participants) | 20 | 3
  Day 36 | 3.3466 [0.9397 to 13.1263] | 0.0385 [0.0385 to 0.0385]
  Day 43: number analyzed (Participants) | 19 | 3
  Day 43 | 5.8947 [1.2107 to 20.2568] | 0.0385 [0.0385 to 0.0385]
  Day 57 | 6.15722 [1.6774 to 18.7678] | 0.0385 [0.0385 to 0.0385]
  Day 180 (Dose 3): number analyzed (Participants) | 19 | 5
  Day 180 (Dose 3) | 3.79298 [1.0944 to 13.2313] | 0.0385 [0.0385 to 0.0385]
  Day 187: number analyzed (Participants) | 18 | 3
  Day 187 | 5.52867 [1.8484 to 23.2002] | 0.0385 [0.0385 to 0.0385]
  Day 194: number analyzed (Participants) | 18 | 3
  Day 194 | 9.62189 [2.7346 to 47.4511] | 0.0385 [0.0385 to 0.0385]
  Day 208: number analyzed (Participants) | 19 | 3
  Day 208 | 11.50262 [2.7182 to 33.0241] | 0.0385 [0.0385 to 0.0385]
  Day 360: number analyzed (Participants) | 17 | 3
  Day 360 | 2.92278 [0.6188 to 11.0412] | 0.05396 [0.0385 to 0.1060]

ADVERSE EVENTS:
Time Frame: Solicited injection site and systemic reactogenicity events were reported from the time of each study vaccination through Day 8 after each study vaccination. Unsolicited non-serious AEs were documented and reported at all visits from signing of the ICF until Day 57, then from Day 180 through Day 208. Serious Adverse Events (SAEs) were collected from the time of the first study vaccination through the last study visit on Day 360.
Arm/Group | HEV-239 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/5
Other Adverse Events (participants affected / at risk) | 19/20 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEV-239 (N=20) | Placebo (N=5)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEV-239 (N=20) | Placebo (N=5)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 7 (12) | 1 (2)
Injection Site Haemorrhage (General disorders) | 2 (3) | 1 (1)
Injection Site Induration (General disorders) | 10 (15) | 1 (1)
Injection Site Pain (General disorders) | 17 (40) | 3 (4)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 5 (7) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 2 (6) | 0 (0)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 11 (18) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT03827395/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03827395/SAP_002.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03827395/ICF_000.pdf